CLINICAL TRIAL: NCT00309855
Title: Mechanisms of Testosterone-Driven Growth-Hormone (GH) Secretion in Aging Men: Modulation of GHRH, GHRP and Somatostatin Action by Estrogenic Versus Androgenic Steroids
Brief Title: Testosterone-Driven Growth-Hormone (GH) Secretion in Aging Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Johannes D. Veldhuis, M.D., Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 319-03
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Aging
MeSH Terms: interventions — Testosterone; Anastrozole; Dutasteride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Double Placebo (Placebo Comparator): (i.m. vehicle 0.5 mL weekly x three injections and oral placebo once daily x 21 days)
  Interventions: Drug: Placebo
- Testosterone IM and oral placebo (Other): IM injections weekly x three injections and oral placebo once daily x 21 days
  Interventions: Drug: Testosterone
- Testosterone and Oral Anastrozole (Other): IM injections weekly x 3 injections and oral daily x 21 days
  Interventions: Drug: Testosterone; Drug: Anastrazole
- Testosterone and Dutasteride (Other): IM injections weekly x 3 injections and oral once daily x 21 days
  Interventions: Drug: Testosterone; Drug: Dutasteride

INTERVENTIONS:
Drug: Placebo — im and orally
  Arms: Double Placebo
Drug: Testosterone — injections
  Arms: Testosterone IM and oral placebo; Testosterone and Dutasteride; Testosterone and Oral Anastrozole
Drug: Anastrazole — orally x 21 days
  Arms: Testosterone and Oral Anastrozole
Drug: Dutasteride — orally x 21 days
  Arms: Testosterone and Dutasteride

SUMMARY:
This study is being done to understand how testosterone, the major male sex hormone, controls the pituitary gland's secretion of growth hormone (GH). GH is an important metabolic hormone, which controls sugar; fat and protein use in the body and maintains muscle strength and bone calcium content. Both testosterone and GH decline in older men. The age-related fall in these hormones probably contributes to relative frailty, reduced quality of life, bone loss, muscle wasting and impaired sexual function.

DETAILED DESCRIPTION:
Repletion of testosterone in older men drives pulsatile GH secretion via conjoint facilitation of feedforward by the primary secretagogues GHRH and GHRP and repression of feedback by the dominant inhibitor, somatostatin; and, in corollary, testosterone acts via aromatization to estradiol and/or reduction to 5 alpha-dihydrotestosterone

ELIGIBILITY:
Inclusion Criteria:

* healthy men between the ages of 50 and 80;
* normal weight (within 30% of ideal body weight defined by New York Metropolitan Life tables); and
* normal hematocrit (greater than 38%);
* community dwelling; and
* voluntarily consenting

Exclusion Criteria:

* recent use of psychotropic or neuroactive drugs (within five biological half-live);
* obesity (outside weight range above);
* anemia (hematocrit < 38%);
* drug or alcohol abuse, psychosis, depression, mania or severe anxiety;
* acute or chronic organ-system disease;
* endocrinopathy, other than primary thyroidal failure receiving replacement;
* nightshift work or recent transmeridian travel (exceeding 3 time zones within 7 days of admission);
* acute weight change (loss or gain of > 2 kg in 6 weeks);
* allergy to administered compounds; and
* unwillingness to provide written informed consent.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Growth Hormone concentration after injections | 24 days
  GH will be measured 4 different times mornings within 16-21 days following the first testosterone injection (day 1).

CONTACTS AND LOCATIONS:
Overall Officials: Johannes D. Veldhuis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States